CLINICAL TRIAL: NCT04958993
Title: A Phase I/II Clinical Study of Anlotinib Hydrochloride Capsule Combined With Concurrent Chemoradiotherapy in the Treatment of Unresectable Stage III Non-small Cell Lung Cancer
Brief Title: A Trial of Anlotinib Combined With Concurrent Chemoradiotherapy in Patients With Unresectable Stage III Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: High incidence of severe radiation pneumonia
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinming Yu, Director of the hospital, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDZLEC2019-069-03
Record Dates: First submitted 2020-08-25; First posted 2021-07-12 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib combined with concurrent chemoradiotherapy (Experimental): Radiotherapy: 1.8-2.0Gy, qd, 54-66Gy, 5 days a week Chemotherapy: squamous cell cancer: paclitaxel + platinum;Adenocarcinoma: pemetrexed + platinum;A cycle of 3W was used, and the appropriate chemotherapy dose was selected by the researcher according to the patient's situation without any restriction on the chemotherapy dose.Pre-induction chemotherapy is allowed.
  Anlotinib: QD, take 2 weeks and stop for 1 week (radiotherapy 1, 2, 4, 5 weeks)
  Interventions: Drug: Anlotinib hydrochloride capsule Combined With Concurrent Chemoradiotherapy

INTERVENTIONS:
Drug: Anlotinib hydrochloride capsule Combined With Concurrent Chemoradiotherapy — radiotherapy (five days a week to accept chest radiotherapy, once per day, every time 1.8-2.0 Gy, total dose 54-66 Gy) AND chemotherapy (Squamous cell carcinoma selective platinum + docetaxel and Adenocarcinoma selective platinum + Pemetrexed) AND Anlotinib Hydrochloride capsule (12mg QD PO d1-14, 21 days per cycle)

SUMMARY:
This is a phase I/II exploratory study to evaluate the efficacy and safety of anlotinib combined with concurrent chemoradiotherapy in the treatment of surgically unresectable stage III non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. The patients volunteered to participate in this study and signed the informed consent;
* 2. Locally advanced (IIIA/IIIC) non-small cell lung cancer patients diagnosed by pathology as newly diagnosed unresectable, inoperable or refused surgery (difficult patients should be evaluated by thoracic multidisciplinary assessment for potential enrollment); .
* 3. Ages 18-75, regardless of gender;
* 4. ECOG score: 0-1;
* 5. Expected survival over 3 months;
* 6. Function of major organs within 7 days prior to treatment meets the following criteria:

A. Standard of blood routine examination (without blood transfusion within 14 days) :

I. Hemoglobin (HB) ≥100 g/L; II. WBC ≥3.0×109/L; Iii. Platelet (PLT) ≥100×109/L.

B. Biochemical examination shall meet the following standards:

I. Total bilirubin (TBIL) ≤1.5 times the upper limit of normal value (ULN); II. AST≤2.5×ULN of alanine aminotransferase (ALT) and aspartate aminotransferase (ASpartate), if accompanied by liver metastasis, ALT and AST≤5×ULN; III. Serum creatinine (Cr) ≤1.5×ULN or creatinine clearance rate (CCr)≥60ml/min; C. Doppler ultrasound evaluation: left ventricular ejection fraction (LVEF) ≥ lower normal limit (50%); D. Pulmonary function assessment: FEV1≥1.45 l/s.

* 7. Patients of childbearing age (including female and female partners of male patients) must take effective birth control measures

Exclusion Criteria:

* 1. Patients who have previously used anlotinib hydrochloride capsules;
* 2. Small cell lung cancer (including mixed small cell and non-small cell cancers);
* 3. Lung squamous cell carcinoma with empty cavity, or non-small cell lung cancer with hemoptysis (> 20ml/day);
* 4. Patients with other malignant tumors other than NSCLC within 5 years before the start of treatment in this study (except those with simple surgical resection and disease-free survival for at least 5 consecutive years, cured cervical carcinoma in situ, cured basal cell carcinoma and bladder epithelial tumor);
* 5. Systemic antitumor therapy, including cytotoxic therapy, signal transduction inhibitors and immunotherapy, is planned within 4 weeks before enrollment or during the medication period of this study.In addition to thymosin, lentinan and other immunomodulator treatment.
* 6. Unmitigated toxicity due to any previous treatment above CTC AE level 1, excluding hair loss;
* 7. Patients with multiple factors affecting oral medication (such as inability to swallow, chronic diarrhea and intestinal obstruction);
* 8. Accompanied by pleural effusion or ascites, causing respiratory syndrome (≥CTC AE level 2 dyspnea);
* 9. Patients with any severe and/or uncontrolled disease, including: A) Patients with unsatisfactory blood pressure control (systolic blood pressure ≥150 mmHg, diastolic blood pressure ≥100 mmHg); B) Having grade I or above myocardial ischemia or infarction, arrhythmia (including QTc ≥480ms), and grade 2 or above congestive heart failure (New York Heart Association (NYHA) classification); C) Active or uncontrolled severe infection (≥CTC AE level 2 infection); D) Antiviral treatment for cirrhosis, decompensated liver disease, active hepatitis or chronic hepatitis; E) Renal failure requires hemodialysis or peritoneal dialysis; F) A history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation; G) poor control of diabetes mellitus (FBG) > 10mmol/L; H) urine routine indicated urinary protein ≥++, and confirmed 24-hour quantitative urinary protein > 1.0g; I) patients with epileptic seizures requiring treatment; J) Patients with gastric ulcer
* 10. Receive major surgical treatment, open biopsy or significant traumatic injury within 28 days before grouping;
* 11. Patients whose tumors have invaded important blood vessels according to imaging findings or whose tumors are likely to invade important blood vessels during the follow-up study according to the judgment of the researchers, resulting in fatal massive hemorrhage;
* 12. Patients with any physical signs or history of bleeding, regardless of severity;Patients with any bleeding or bleeding event ≥CTCAE level 3 within 4 weeks prior to enrollment have unhealed wounds, ulcers or fractures;
* 13. Occurrence of ARTERIAL/venous thrombotic events, such as cerebrovascular accidents (including temporary ischemic attacks), deep venous thrombosis and pulmonary embolism within 6 months;
* 14. Persons with a history of abuse of psychotropic substances and who cannot be cured or have mental disorders;
* 15. Pregnant and lactating women;
* 16. Participated in other clinical trials of anti-tumor drugs within 4 weeks;
* 17. The researcher considered that there were other conditions that were not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2021-11-22 (Actual)

PRIMARY OUTCOMES:
Progress free survival (PFS) for phase Ⅱ | up to 30 months
  PFS defined as the time from first dose of study treatment until the first date of either objective disease progression or death due to any cause.
Maximum Tolerance Dose (MTD) for phaseⅠ | From enrollment to completion of study. Estimated about 18months
  Maximum Tolerance Dose (MTD) is the dose of treatment in the cohort where there are 2 cases of DLT reported.Dose Limiting Toxicity (DLT) is referred to grade 3 non-hematological toxicity or grade 4 hematological toxicity according to NCI CTCAE 5.0 criteria

SECONDARY OUTCOMES:
Overall Survival (OS) | From randomization until death (up to 30 months)
  OS is defined as the time until death due to any cause.
Objective Response Rate (ORR) | each 42 days up to intolerance the toxicity or PD (up to30 months)
  ORR is defined as the percentage of subjects with evidence of a confirmed complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1.prior to progression or any further therapy.

CONTACTS AND LOCATIONS:
Overall Officials: JINGMIN YU, PhD, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Shandong Cancer Hospital, Jinan, Shandong, China